CLINICAL TRIAL: NCT03905252
Title: Biomarkers for Human Heart Failure
Acronym: Biomarkers
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John C Burnett, Principal Investigator, Mayo Clinic
Other Study IDs: IRB # 09-003156
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: CHF

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — : Single blood draw, random urine and 24-hr urine collection
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: sample analysis — blood, Random urine sample and 24-hour urine samples

SUMMARY:
The purpose of this study is to establish the various ranges of proteins that can be assayed in the plasma and urine from hospitalized patients with all classes of heart failure and/or STEMI (ST-segment elevation myocardial infarction)/NSTEMI (Non-ST-segment elevation myocardial infarction), as well as history reviews.

DETAILED DESCRIPTION:
Schematic Design of the Study: Single blood draw, one random urine and 24-hr urine collection from hospitalized patients with chronic/acute heart failure and/or STEMI-NSTEMI. If there should be a subsequent hospitalization,another collection of a 45 ml blood sample, random urine and one 24-hour urine collection may be completed if indicated at initial hospitalization.

Aims:

The purpose of this study is to attempt to establish the various ranges of proteins that can be assayed from the plasma and urine of patients with all classes of heart failure and MI (myocardial infarction). Follow-up hospitalizations may result in another 45 ml blood draw, random urine and 24-hr. urine collection to evaluate the outcome of the heart failure treatment used with the previous hospitalization, if indicated in consent. A history review will be necessary as well.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosis of Acute decompensated heart failure

Exclusion Criteria:

• Hemoglobin less than 10, active cancer, or amyloidosis Patient with dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eight Hundred HF patients hospitalized for symptomatic HF at Mayo Clinic Hospital - St Mary's Campus, Rochester, Minnesota
Sampling Method: Non-Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2024-02 (Actual); Study Completion 2024-02 (Actual)

PRIMARY OUTCOMES:
uAGT levels in high-risk chronic HF patients | 10 years
  This study will provide new knowledge of the pathology and outcomes predicted by the use of uAGT in symptomatic chronic HF patients at high risk for future hospitalization and death.
Natriuretic peptide levels in ADHF patients | 20 years
  new knowledge of pathology and outcomes in ADHF patients

CONTACTS AND LOCATIONS:
Overall Officials: John C Burnett, M.D., Principal Investigator — Mayo Foundation
Locations (1):
- Mayo Foundation, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No